CLINICAL TRIAL: NCT05935111
Title: Obesity and Physical Activity: Feasibility Study
Brief Title: Physical Activity: Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Binghamton University (Other)
Collaborators: Lehigh University (Other); Ascension Health (Industry)
Responsible Party: Principal Investigator, Seungmin Lee, Assistant Professor, Binghamton University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: RNY20230009
Record Dates: First submitted 2023-06-27; First posted 2023-07-07 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Obesity; Physical Activity; Self-efficacy; Online Intervention; Accelerometers
Keywords: obesity; physical activity; self-efficacy; information and communication technology; accelerometers
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity Self-efficacy (PAS) group (Active Comparator): Participants assigned to the PAS group will proceed through the weight management program provided by the center and will be given 4 weeks of 24-hour access to the PAS intervention during data collection for this study. The login credential for PAS participants will provide access to both the PAS intervention and to a secure website to complete data collection at W1, W2, and W3.
  Interventions: Behavioral: Physical Activity Self-efficacy (PAS) intervention
- Usual Care (UC) group (No Intervention): Participants assigned to the UC group will proceed through the weight management program provided by the center. The login credential for UC participants will provide access to a secure website to complete data collection (i.e., a survey battery, physical activity monitoring) at W1, W2, and W3.

INTERVENTIONS:
Behavioral: Physical Activity Self-efficacy (PAS) intervention — The PAS intervention will be a web-based intervention to address the unique barriers to physical activity in adults with obesity, based on self-efficacy theory and effective behavioral change techniques. Self-efficacy is specified as a mediating psychological variable in the conceptual model for the promotion of physical activity. Self-efficacy refers to domain-specific beliefs (e.g., job-, transport-, domestic-, leisure-related physical activity) about their ability to execute differing levels of performance given situational demands. There is a rich literature on the importance of targeting self-efficacy as a modifiable mediating variable in PA-promoting interventions. Also, the PAS intervention will consist of effective behavioral change techniques (e.g., action planning, teach to use prompts/cues, goal setting, etc.).
  Other Names: PAS intervention
  Arms: Physical Activity Self-efficacy (PAS) group

SUMMARY:
The Physical Activity Self-efficacy (PAS) intervention is a web-based behavioral intervention newly developed to promote physical activity in adults with obesity. The conceptual framework for the PAS intervention is based on self-efficacy theory. The objective of this study is to investigate the feasibility and acceptability of implementing the PAS online intervention for adults with obesity recruited from a local weight management center in the United States of America (USA). The study design is a prospective, double-blind, parallel group randomized pilot trial. Thirty participants will be randomly assigned to the PAS group or usual care group to achieve a 1:1 group assignment. Recruitment of participants is scheduled to begin in January 2024 or earlier at a local weight management center within a private healthcare system in the USA. There are five eligibility criteria for participation in this study (e.g., a body mass index ≥ 25.00 kg/m2). Eligibility verification and data collection will be conducted online. Three waves of data collection will take up to 14 weeks depending on participants' progress in the study. Instruments designed to measure demographic information, anthropometric characteristics, self-efficacy, and acceptability will be included in the survey battery. A research-grade accelerometer will be used to measure free-living physical activity objectively. Data will be analyzed using descriptive statistics and inferential statistical models under an intention-to-treat approach. This study will be sponsored by the Transdisciplinary Areas of Excellence Seed Grant Program from Binghamton University.

ELIGIBILITY:
There are five eligibility criteria for participation in this study. Values for each of the eligibility criteria will be based on self-report by the potential participant. Potential participants who do not meet one or more of the eligibility criteria will be informed that they are ineligible for the study and then will be taken to the exit page from the PAS website (http://pasintervention.com/login).

* The first criterion is being between 18 and 64 years old, consistent with evidence-based age groupings for global recommendations on physical activity for health.
* The second criterion is a body mass index (BMI) ≥ 25.00 kg/m2, consistent with many physical activity interventions in adults with obesity. A justification for this criterion is the need to promote physical activity in a BMI-based population in which few individuals may meet public health guidelines for physical activity.
* The third criterion is the ability to access the online intervention. This criterion will be assessed by asking them to confirm that they will have access to a technological device (e.g., computer, smart phone) that can access the online intervention via a web browser.
* The fourth criterion is a willingness to comply with instructions for physical activity monitoring. This criterion will be assessed by asking them if they are willing to wear a physical activity monitor on their waist for two 7-day intervals and complete a daily log sheet regarding wear time during each of the two 7-day intervals in the study. A justification for this criterion is based on previous studies where a similar question was asked to potential participants at screening. Those who indicate a willingness to comply with instructions for physical activity monitoring will be asked to provide information about their non-dominant hand.
* The final criterion is a willingness to respond to study-related contacts (e.g., email, text message, phone call). A justification for this criterion is that participants will be asked to complete some tasks in a specifically structured schedule.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — What is your gender?
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the feasibility of implementing the PAS intervention (e.g., recruitment rate, eligibility rate) for adults with obesity recruited from a local weight management center in the USA. | By Week 7
  The feasibility of implementing the PAS online intervention for adults with obesity recruited from a local weight management center in the USA will be assessed with descriptive statistics. Descriptive statistics will include (a) recruitment rate, (b) eligibility rate, (c) consent rate, (d) participation rates, and (e) retention rates.
the acceptability of implementing the PAS intervention (e.g., engagement, accelerometer-based assessment of physical activity) for adults with obesity recruited from a local weight management center in the USA. | By Week 7
  The acceptability of implementing the PAS online intervention for adults with obesity recruited from a local weight management center in the USA will be assessed with descriptive statistics. Descriptive statistics will include acceptability of the PAS intervention (e.g., engagement behavior, subjective experience) and acceptability of accelerometer-based assessment of physical activity.
a preliminary effect size estimate for each direct effect depicted in the conceptual model for the PAS online intervention. | By Week 14
  Within 7 days after the W1 and W3 survey battery, participants will be asked to enter a code into the PAS intervention website in order to start wearing a physical activity monitor for the next consecutive 7 days. They will be instructed to wear a research-grade accelerometer, ActiGraph wGT3X-BT, on their waist.
  The primary measure of physical activity in this study will be the average minutes per day of Moderate to Vigorous Physical Activity (MVPA) based on both widely accepted recommendations for health-enhancing physical activity. Instruments designed to measure the acceptability of accelerometer-based assessment of physical activity and self-reported physical activity will also be included in the W1 and W3 physical activity monitoring.

SECONDARY OUTCOMES:
Self-efficacy to engage | By Week 7
  After completion of the introductory challenges, PAS participants will be asked at W2 to respond to the following item: How confident are you in your current ability to get yourself to complete at least 24 post-introductory challenges within the next four weeks?
Physical activity self-efficacy | By Week 3, By Week 7, By Week 14
  Physical activity self-efficacy will be measured from participants at W1, W2, and W3 with the physical activity self-efficacy scale. The 48-item scale is a modified version of the exercise self-efficacy scale.
Self-efficacy to regulate physical activity | By Week 3, By Week 7, By Week 14
  Self-efficacy to regulate physical activity will be measured from participants at W1, W2, and W3 with the self-efficacy to regulate physical activity scale. The 13-item scale is a modified version of the barriers self-efficacy scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Guthrie, Binghamton, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Participants will be asked to provide some personally identifiable information (e.g., phone number) during enrollment in the study. This personally identifiable information and all other data collected online (e.g., online survey battery) will be collected via a secure website maintained by authorized research staff employed by Lehigh University. The research staff will share all data collected via the secure website with authorized research staff employed by Binghamton University. All data collected will be kept confidential to the maximum extent allowable by law. Data obtained from this research will be stored in such a way that human participants cannot be identified. Specifically, all account holders will be assigned a coded identification number in the stored data. The list connecting each participant with an identification number will be kept protected, encrypted, private, and only accessible to authorized research staff at Lehigh University and Binghamton University.
Supporting Information: Study Protocol, ICF
Time Frame: 10/02/2023 - 12/31/2024
Access Criteria: authorized research staff employed by Lehigh University and Binghamton University
URL: http://pasintervention.com/login

REFERENCES:
- [Derived] Lee S, Lahoda K, Myers N, Horowitz A, Freeland M, Einav E, Buckingham-Schutt L, Welk G. Initial outcomes from the Confident Moves online intervention to promote physical activity in adults with obesity: a longitudinal feasibility and acceptability pilot trial. BMC Public Health. 2025 Oct 13;25(1):3466. doi: 10.1186/s12889-025-24763-0. PMID 41083971
- [Derived] Lee S, Lahoda K, Myers ND, Horowitz A, Chiu K, Begdache L, Einav E. Physical activity self-efficacy online intervention for adults with obesity: protocol for a feasibility study. Pilot Feasibility Stud. 2024 Feb 26;10(1):40. doi: 10.1186/s40814-024-01468-6. PMID 38409075